CLINICAL TRIAL: NCT05050344
Title: Descriptive Bicentric Study of Moya Moya Syndrome and Disease in Sickle Cell Disease Patients and Not Sickle Cell Disease
Brief Title: Moya Moya Syndrome With or Withtout Sickle Cell Disease
Acronym: BMM-ScD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL21_0343
Record Dates: First submitted 2021-06-10; First posted 2021-09-20 (Actual); Last update posted 2021-09-24 (Actual); Status verified 2021-06

CONDITIONS: Moya Moya Disease
Keywords: Moya Moya syndrome; Moya Moya
MeSH Terms: conditions — Moyamoya Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Moya Moya disease or syndrome ar characterized by a progressive or occlusion of the intracranial carotid arteries and their mainproximal branches, followed by the development of fragile neovessels at the base of the skull, leding to a high risk of both ischemic and hemorragic stroke over time. Moya Moya syndrome are associated to a variety of disease, which main frequent is sickle cell disease (SCD).

Among patients with SCD who had suffered from at least one ischemic stroke, the prevalence of moya moya syndrome was estimated up to 43%. In general, therapeutic strategies in Moya Moya to prevent first ever ou recurrent stroke can be divided into conservative medical treatment and surgical revascularisation (direct bypass, indirect bypass or combined bypass).

The aim of this study is to compare prognosis of patients with Moya Moya syndrome associated with sickle cell disease or not. The investigators retrospectiveluy analysed medical chart from 2010 to 2021 of patients with Moya Moya disease or syndrome at two French university hospitals (including a center of the french West Indies where prevalence of sickle cell disease is high). The diagnosis was based on angiography or MRI records showing uni- or bilateral stenosis of distal intracranial internal carotide arteries or middle cerebral arteries associated wirh classic collateral network.

Main endpoint will be comparison of a composite outcome defined as time from Moya Moya diagnosis to first or recurrent stroke or bad prognosis achivement (defined by modified Rankin score >2)

ELIGIBILITY:
Inclusion criteria:

* age >=15
* patients at diagnosis of Moya Moya disease and syndrome

Exclusion criteria:

* misclassified patients
* clinical diagnosis of MM not confirmed by angiography or MRI

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients >=15 years of age at diagnosis of Moya Moya disease and syndrome from january 2010 to february 2021 at Montpellier and Martinique University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-05-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
time from Moya Moya diagnosis to first or recurrent stroke or bad prognosis achivement | 1 day
  composite endpoint of outcome defined as time from Moya Moya diagnosis to first or recurrent stroke or bad prognosis achivement (defined by modified Rankin score >2)

SECONDARY OUTCOMES:
Time from MM diagnosis to Stroke | 1 day
  Time from MM diagnosis to Stroke
poor prognosis or death | 1 day
  poor prognosis or death (mRS> 2) at the last clinical evaluation.

CONTACTS AND LOCATIONS:
Overall Officials: Estelle BRITHMER, Resident, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC